CLINICAL TRIAL: NCT00001587
Title: A Phase I Study of Isolated Hepatic Portal and Arterial Perfusion (IHP) With Escalating Dose Melphalan for Primary or Metastatic Unresectable Cancers of the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970200; 97-C-0200
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Liver Neoplasms; Neoplasm Metastasis
Keywords: Hyperthermia; Metastases; Organ Perfusion; Regional Therapy
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Hyperthermia | interventions — Melphalan

INTERVENTIONS:
Procedure: Isolated hepatic portal and arterial perfusion
Drug: Melphalan

SUMMARY:
Patients with unresectable primary or metastatic cancer confined to the liver will undergo a 1 hour hyperthermic isolated hepatic perfusion (IHP) via the portal vein and hepatic artery with escalating dose melphalan. Patients eligible for this protocol are those with non-colorectal histologies and those with colorectal cancer previously treated with intra-arterial FUDR. Hepatic and systemic toxicity, response to treatment, duration of response, and survival will be followed.

DETAILED DESCRIPTION:
Patients with unresectable primary or metastatic cancer confined to the liver will undergo a 1 hour hyperthermic isolated hepatic perfusion (IHP) via the portal vein and hepatic artery with escalating dose melphalan. Patients eligible for this protocol are those with non-colorectal histologies and those with colorectal cancer previously treated with intra-arterial FUDR. Hepatic and systemic toxicity, response to treatment, duration of response, and survival will be followed.

ELIGIBILITY:
Histologically or cytologically proven measurable primary or metastatic non-colorectal cancer limited to the parenchyma of the liver with no evidence of unresectable extrahepatic disease by preoperative radiological studies.

Limited resectable extrahepatic disease is acceptable.

Patients with colorectal cancer previously treated with intrahepatic arterial infusional therapy using FUDR, those with aberrant arterial anatomy such that infusional therapy is not possible, or those with limited extrahepatic disease such that regional therapy is not indicated will be eligible for this protocol.

Patients must have had no chemotherapy, radiotherapy, or biologic therapy for their malignancy in the month prior to the liver perfusion and must have recovered from all side effects.

Patients must have an ECOG performance standard of 0, 1 or 2 on the day prior to treatment.

Patients must have adequate hepatic function as evidence by bilirubin less than 2.0 and a PT and PTT that are within 1-2 seconds of the upper normal limit.

No patients with biopsy proven cirrhosis or evidence of significant portal hypertension by history, endoscopy, or radiologic studies will be included.

No patients with a history of congestive heart failure with an LVEF of equal to or less than 40% will be included.

No patients with COPD or other chronic pulmonary disease with PFT's less than 50% predicted for age will be included.

Patients must be 18 years of age or older.

Patients must have a platelet count greater than 100,000, a HCT greater than 27.0, a white blood count greater than 3000/ micrograms, and a creatinine less than or equal to 1.5 or a creatinine clearance of greater than 60 ml/min.

No pregnant patients or nursing mothers will be eligible.

Patients must not be taking immunosuppressive drugs or on chronic anticoagulation.

Patients must not have an active infection.

Patients with severe allergic reactions to iodine contrast which can not be controlled by premedication with antihistamines and steroids are not eligible as a hepatic angiogram is needed for this procedure.

Patients must not have HIV disease.

Patients must be aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks.

The patient must be willing to sign an informed consent.

Patients must not have a history of veno occlusive disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1997-09; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Alexander HR Jr, Bartlett DL, Libutti SK. Isolated hepatic perfusion: a potentially effective treatment for patients with metastatic or primary cancers confined to the liver. Cancer J Sci Am. 1998 Jan-Feb;4(1):2-11. No abstract available. PMID 9467038
- [Background] Alexander HR Jr, Bartlett DL, Libutti SK, Fraker DL, Moser T, Rosenberg SA. Isolated hepatic perfusion with tumor necrosis factor and melphalan for unresectable cancers confined to the liver. J Clin Oncol. 1998 Apr;16(4):1479-89. doi: 10.1200/JCO.1998.16.4.1479. PMID 9552055